CLINICAL TRIAL: NCT01469676
Title: Effects of CPB-leukocyte Filtration on Interleukins Serum Levels and Pulmonary Function.
Brief Title: Effects of Cardiopulmonary Bypass (CPB)-Leukocyte Filtration on Interleukins Serum Levels and Pulmonary Function
Acronym: PulmFunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: InCor Heart Institute (Other); Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Maria José Carvalho Carmona, Effects of CPB-leukocyte Filtration on Interleukins Serum Levels and Pulmonary Function, University of Sao Paulo
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: Leukocyte Filtration
Record Dates: First submitted 2011-06-22; First posted 2011-11-10 (Estimated); Last update posted 2011-11-10 (Estimated); Status verified 2011-11

CONDITIONS: Systemic Inflammatory Response Syndrome (SIRS); Leukocyte Disorders; Complications Due to Coronary Artery Bypass Graft
Keywords: Coronary Artery Bypass Surgery; Cardiopulmonary Bypass; Leukocyte Reduction Filtrations; Pulmonary Function; Systemic Inflammatory Response
MeSH Terms: conditions — Systemic Inflammatory Response Syndrome; Leukocyte Disorders | interventions — Leukocyte Reduction Procedures

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (No Intervention): In the Control group, a standard arterial line filter was inserted on CPB circuit.
- Filtering Group (Experimental): In the Filtering group, a leukocyte filter was inserted in the arterial line circuit.
  Interventions: Device: Filtering group LG-6, Pall Biomedical Products

INTERVENTIONS:
Device: Filtering group LG-6, Pall Biomedical Products — In Filtering group, a Leukocyte filter (LG-6, Pall Biomedical Products) was placed on the CPB arterial line circuit, trying to filter the white blood cells.
  Other Names: LeukoGard-6; Leukocyte depletion; Leukoreduction
  Arms: Filtering Group

SUMMARY:
To test the hypothesis that leukocyte filtering during cardiopulmonary bypass (CPB) might reduce the inflammatory response and protect the lungs against the acute injury

DETAILED DESCRIPTION:
BACKGROUND AND OBJECTIVES: The extension of the systemic inflammatory response observed after cardiopulmonary bypass (CPB) in cardiac surgery is associated to postoperative pulmonary dysfunction degree. The leukocyte depletion during CPB can modify that response. The aim of this study was to evaluate the effects of leukocyte filtering on the inflammatory response and lung function in patients undergoing coronary artery bypass grafting.

METHODS: After approval by the institutional ethical committee, a prospective randomized study was performed to compare nine patients undergoing coronary artery bypass grafting (CABG) using leukocyte filtration in the arterial line (LG-6, Pall Biomedical Products) and eleven others submitted to standard CPB. Chest CT, oxygenation analysis and a complete leucocyte count were performed before surgery. After intravenous anesthesia induction, patients were mechanically ventilated with tidal volume of 8 mL.kg-1, with FiO2 0.6, and PEEP of 5 cm H2O, except during CPB. Haemodynamic data, PaO2/FiO2, shunt fraction, interleukins, elastase and myeloperoxidase were evaluated before and after CPB, at the end of surgery, 6, 12 and 24 hours after surgery. Chest CT was repeated on the first postoperative day. Data were analyzed using two-factor ANOVA for repeated measures.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing coronary artery bypass grafting (CABG), having their physical state classified as PII and PIII, according to the American Society of Anesthesiologists (ASA). Surgical risk was stratified according to Parsonnet criteria, and only patients considered low to moderate risk were admitted.

Exclusion Criteria:

* Subjects older than 70 years
* Body mass index (BMI) over 35 kg/m2
* Congestive heart failure (CHF) greater than class III (NYHA)
* Left ventricle ejection fraction less than 40%
* Submitted to recent surgery
* creatinine ≥ 1.4 mg / dL or in use of oral anticoagulants were excluded

Max Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2007-02; Primary Completion 2010-02 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Effects of CPB-leukocyte Filtration on Interleukins Serum Levels and Pulmonary Function. | 24 hours
  The primary outcome was the evaluation of the effects of leukocyte filtration on lung function in patients undergoing coronary surgery.

SECONDARY OUTCOMES:
Evaluation of the effects of leukocyte filtration on the inflammatory response in patients undergoing coronary surgery. | 24 hours
  The secondary outcome was the evaluation of the effects of leukocyte filtration on the inflammatory response in patients undergoing coronary surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Maria José C Carmona, phd, Principal Investigator — U Sao Paulo